CLINICAL TRIAL: NCT07316738
Title: Effect of Ozonated Gel Phonophoresis on Pain and Functional Disability in Patients With Chronic Supraspinatus Tendinitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohsen Ali Abdallah, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/006041
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Supraspinatus Tendinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozonated gel phonophoresis + conventional treatment (Experimental): Twenty patients will receive ozonated gel phonophoresis in addition to conventional treatment, three times per week for four weeks.
  Interventions: Other: ozonated gel phonophoresis; Other: conventional treatment
- conventional treatment (Active Comparator): Twenty patients will receive conventional treatment consisting of hot pack application and stretching exercises targeting the upper trapezius and pectoralis minor muscles. Stretching will be performed for three repetitions, each held for 30 seconds with 30 seconds of rest between repetitions. This will be followed by strengthening exercises for the external shoulder rotators, lower trapezius, and serratus anterior muscles using color-coded elastic resistance bands, performed as three sets of ten repetitions for each muscle group. In addition, ultrasound therapy will be applied at a frequency of 1 MHz and an intensity of 0.8 W/cm² for 7 minutes. Treatment sessions will be conducted three times per week for four weeks.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: ozonated gel phonophoresis — Patients will receive ultrasonic with ozonated gel as a coupling medium (phonophoresis) (1 MHz, 1 W/cm2 continuous mode) for 5 min, three times per week for four weeks.
  Arms: ozonated gel phonophoresis + conventional treatment
Other: conventional treatment — Patients will receive conventional treatment consisting of hot pack application and stretching exercises targeting the upper trapezius and pectoralis minor muscles. Stretching will be performed for three repetitions, each held for 30 seconds with 30 seconds of rest between repetitions. This will be followed by strengthening exercises for the external shoulder rotators, lower trapezius, and serratus anterior muscles using color-coded elastic resistance bands, performed as three sets of ten repetitions for each muscle group.Treatment sessions will be conducted three times per week for four weeks.

SUMMARY:
This study will be conducted to investigate the effect of ozonated gel phonophoresis on pain intensity, shoulder joint range of motion, and functional disability in patients with chronic supraspinatus tendinitis grades I and II.

DETAILED DESCRIPTION:
Tendinopathy is a condition in which pain arises on tendon near origin or insertion due to repetitive activities and reduced functional level, it occurs when the tendon does not properly heal.

Thirty percentages of tendinopathies in musculoskeletal conditions are shoulder pain related where supraspinatus tendinitis is the third most prevalent problem.

The primary function of the supraspinatus muscle is shoulder abduction, particularly movements that elevate the arm overhead. During these motions, the supraspinatus tendon repeatedly passes beneath the acromion process of the scapula, which can result in impingement and subsequent inflammation. If this condition progresses, an unexpected force or trauma may cause partial or complete rupture of the tendon.

Phonophoresis was first used to treat polyarthritis of hand by driving hydrocortisone ointment into inflamed areas in 1994. Since then it has been used in the treatment of various dermatological and musculoskeletal disorders.

The major medications used today with phonophoresis include the anti-inflammatories (cortisol, dexamethasone, salicylates) and local anaesthetics (lidocaine). Cameroy reports success using Carbocaine phonophoresis before closed reduction of Colles fractures.

The main purpose of phonophoresis is to achieve a suitable and fast concentration of drug in the tissue without inactivating the drug molecules with no side effects. In this efficient method, this has had wide utility in physical therapy and sports medicine. The drug is applied locally at the target site and messaged with a therapeutic ultrasound applicator.

Ozone therapy is a potential minimally invasive, conservative treatment that can be used alone or in conjunction with other therapies to help people with musculoskeletal diseases perform better and experience less pain. According to various studies, the effectiveness and safety of ozone therapy have primarily been researched in cases of knee osteoarthritis and on back pain.

Several papers suggested relevant medical features of O3, including inflammatory modulation and circulatory stimulation, with multiple applications in several medical fields including wound healing, ischemic disorders, infections and chronic inflammatory conditions like musculoskeletal disorders.

In the available literature there is no studies were done to identify the effect of ozonated gel phonophoresis in management of patients with chronic supraspinatus tendinitis grade I & II.

So this study may add a piece of information to the therapists in the governmental hospitals and private clinics to be aware about the efficacy of this approach during dealing with patients of chronic supraspinatus tendinitis grade I & II.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 30-60 years old from both genders.
* The patients will be assigned to the study will be diagnosed with grade I or II supraspinatus tendinitis based on Neer's classification.
* The patients suffered from supraspinatus tendinitis for more than 3 months and taking non-steroidal anti-inflammatory drugs suggested by orthopedist.
* All patients have body mass index between 18.5 and 29.9 kg/m2.

Exclusion Criteria:

* Grades III of supraspinatus tendinitis. (Bone spurs and tendon rapture)
* Any past shoulder surgical interventions. (Rotator cuff repair, labrum tear and open reduction internal fixation)
* Shoulder joint instability
* Shoulder fracture.
* Non-cooperative subjects.
* Neuromuscular diseases (spinal muscular atrophy, whiplash injury)
* Cardiovascular disease.
* History of cancer.
* Systemic diseases such as rheumatoid arthritis, Reiter's syndrome, or diabetes.
* Severe medical and neurological or psychiatric disorders.
* Pregnant and lactating women.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain intensity of shoulder joint | 4 weeks
  Pain intensity of the shoulder joint will be assessed using the Visual Analog Scale (VAS) in patients with chronic supraspinatus tendinitis. Patients will be asked to place a mark on a horizontal line to indicate the intensity of their pain, where the left end represents no pain and the right end represents the worst pain imaginable. VAS scores will be interpreted as follows: 0-30 indicates mild symptoms, 31-60 indicates moderate symptoms, and 61-100 indicates severe symptoms.
Assessment of Functional disability | 4 weeks
  The Quick Disabilities of the Arm, Shoulder, and Hand Scale (Quick DASH; Q-DASH) will be used to evaluate shoulder dysfunction. The QuickDASH consists of 11 items extracted from the original 30-item DASH questionnaire, including 8 function/disability items and 3 symptom items. Each item is scored on a 5-point scale ranging from 1 (no difficulty) to 5 (unable to do), with total scores ranging from 0 to 100, where higher scores indicate greater disability.

SECONDARY OUTCOMES:
Assessment of Shoulder abduction range of motion | 4 weeks
  A digital goniometer will be used to assess shoulder joint abduction range of motion in patients with chronic supraspinatus tendinitis before and after the treatment sessions. Measurements will be taken with the patient in the supine position. The fulcrum of the goniometer will be centered at the anterior aspect of the acromion process, the stationary arm will be aligned parallel to the midline of the torso, and the moving arm will be aligned with the midline of the humerus, pointing toward the medial epicondyle of the elbow.
Assessment of Shoulder External Rotation range of motion | 4 weeks
  Shoulder joint external rotation range of motion will also be assessed using a digital goniometer before and after the treatment sessions in patients with chronic supraspinatus tendinitis. The patient will be positioned supine during measurement. The fulcrum of the goniometer will be centered over the olecranon process of the elbow, the stationary arm will be aligned perpendicular to the floor, and the moving arm will be aligned with the ulna, pointing toward the ulnar styloid process.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ramzy Lasheen, PhD, Study Chair — Assistant Professor, Cairo University; Nouran Ahmed Ibrahim, PhD, Study Director — Lecturer, Cairo university; Mohamed Osama Hegazy, PhD, Study Director — Professor, Banha University
Locations (1):
- AL-Nasaem outpatient clinic, Cairo, Egypt